CLINICAL TRIAL: NCT01293916
Title: Spica Casting in Pediatric Femur Fractures: A Prospective Randomized Controlled Study of Single Leg vs Double Leg Spica Casts
Brief Title: Spica Casting in Pediatric Femur Fractures: Study of Single Leg Versus Double Leg Spica Casts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00005452
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Femur Fracture
Keywords: pediatric; femur; femoral; fracture; spica; cast; diaphyseal; single; double; patient age 2 to 6 years old
MeSH Terms: conditions — Femoral Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double leg spica cast (Active Comparator): The current accepted treatment is the double leg spica cast in the treatment of pediatric diaphyseal femur fractures.
  Interventions: Other: Spica casting
- Single leg spica casts (Experimental): The study group is the single leg spica cast group
  Interventions: Other: Spica casting

INTERVENTIONS:
Other: Spica casting — single versus double leg spica casting

SUMMARY:
Prospective randomized controlled trial comparing use of single leg spica with double leg spica casts in the treatment of pediatric femur fractures in children ages 2 through 6 years old.

DETAILED DESCRIPTION:
Introduction

* double-leg spica casting is the treatment of choice at many centers for the treatment of diaphyseal femur fractures in children 2 to 6 years old.
* Investigators hypothesize that these patients can be effectively treated with single-leg spica casting and that such treatment will result in easier care and better patient function during treatment.

Methods

* Prospective randomized controlled study of patients between 2 and 6 years old with diaphyseal femur fractures
* patients randomly assigned to either immediate single or double-leg spica casting groups after consent was obtained
* Radiographs serially evaluated for maintenance of reduction with respect to length, varus/valgus angulation and procurvatum/recurvatum angulation
* After casts removal, the Activity Scale for Kids (Performance Version) questionnaire and a custom written survey were given to parents evaluating ease of care and function of children during treatment.

ELIGIBILITY:
Inclusion Criteria:

* diaphyseal femur fracture
* age between 2 and 6 years old

Exclusion Criteria:

* underlying bone disorder
* neuromuscular disease

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Acceptable fracture healing | 8 weeks
  evaluation of shortening, angulation, and rotation radiographically at time of fracture healing

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Leu, MD, Study Director — Johns Hopkins University; Paul D Sponseller, MD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States